CLINICAL TRIAL: NCT04362241
Title: DEXTENZA VS. PREDNISOLONE ACETATE 1% in the Incidence of Pseudophakic Macular Edema in Patients With Diabetic Retinopathy Undergoing Cataract Surgery
Brief Title: DEXTENZA VS. PREDNISOLONE ACETATE 1% Macular Edema With Diabetic Retinopathy After Cataract Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ophthalmic Consultants of the Capital Region (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OphthalmicConsultantsOC
Record Dates: First submitted 2020-04-10; First posted 2020-04-24 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Retinopathy, Diabetic
MeSH Terms: conditions — Diabetic Retinopathy | interventions — prednisolone acetate

STUDY DESIGN:
Intervention Model Description: This prospective study will use a fellow-eye design for 30 participants, summing to 60 eyes total. All eyes will receive cataract surgery. Per participant, one eye will be randomized to receive DEXTENZA® insertion at the end of the surgery, while the other eye will be assigned to a standard of care prednisolone acetate 1% eye drop regimen.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dextenza (Experimental): Sustained release Dexamethasone 0.4mg
  Interventions: Drug: Prednisolone Acetate 1% Ophthalmic Suspension [PRED FORTE]
- Prednisolone Acetate 1% (Active Comparator): Prednisolone Acetate Ophthalmic drops
  Interventions: Drug: Prednisolone Acetate 1% Ophthalmic Suspension [PRED FORTE]

INTERVENTIONS:
Drug: Prednisolone Acetate 1% Ophthalmic Suspension [PRED FORTE] — Prednisolone Acetate 1% ophthalmic drops
  Other Names: Prednisolone Acetate 1%

SUMMARY:
The complicated schedules for administering topical steroid eye drops combined with forgetfulness and physical difficulties instilling the drops may compromise compliance; which in turn could increase the risk for secondary complications such as PME post-cataract surgery, especially in a high-risk diabetic population. Dextenza, a sustained- release steroid insert, could help preclude adherence difficulties and provide better bioavailability, being as effective as, or more effective than steroid drops in preventing PME. The aim of this study is to assess the incidence of PME in diabetic patients undergoing cataract surgery when comparing the Dextenza insert to topical prednisolone acetate 1% drops.

DETAILED DESCRIPTION:
This prospective, open-label, single-center, randomized, fellow-eye, investigator-sponsored clinical study seeks to investigate the incidence of PME in diabetic patients with any level of background diabetic retinopathy undergoing cataract surgery treated with a 0.4mg dexamethasone intracanalicular insert when compared to standard of care prednisolone acetate 1% QID/1 week, TID/ 1 week, BID/ 1 week, QD/1 week. Topical NSAIDs will not be used in this study and all patients will receive an intracameral injection of moxifloxacin at the end of the surgical procedure. After screening a patient for inclusion and exclusion criteria, and gaining informed consent, each eye will undergo cataract surgery on separate days. The second eye will be operated on within 60 days of the first eye's surgery. One eye will be randomized to receive the dexamethasone insert using a coin flip. The other eye will be prescribed a prednisolone acetate 0.1% eye drop QID/ 1 week, TID/ 1 week, BID/1 week, QD/ 1 week regimen. The dexamethasone insert will be placed 2-4 days before surgery (Day -4 to Day-2) and those randomized to receive prednisolone acetate will start 2-4 days before surgery. After surgery, each eye will be followed for a period of approximately 60 days, consisting of four post-op follow-up visits (eight total post-op visits per patient). Primary and secondary endpoints will be assessed alongside standard-of-care procedures at all study visits . Adjusting for the enrollment period, the study will last a total of approximately 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Binocular
* >18 years old
* Any level of Background Diabetic Retinopathy
* Cataract surgery candidate in each eye
* Pre-operative OCT and Fluorescein Angiography showing no Macular edema

Exclusion Criteria:

* Participant cannot complete second eye operation within 60 days of the first cataract surgery
* Maintains regular use of systemic or ocular steroids at time of enrollment
* Maintains regular use of systemic or ocular non-steroidal anti-inflammatory drugs at time of enrollment
* Anterior chamber cells present at time of enrollment
* Recent febrile illness that precludes or delays participation for 90 days
* Pregnancy or lactation
* Known allergy to dexamethasone
* Known allergy to prednisolone
* Preexisting retinal disease including uveitis, nondiabetic retinal disease, choroidal disorders, diabetic macular edema.
* Posterior capsule rupture or other intraoperative complication in first eye operated on
* Amblyopia
* Anti-VEGF injections within 6 months prior to surgery day.
* Intraocular steroid injection within 6 months prior to surgery day.
* Intraocular surgeries within 6 months prior to surgery day.
* Laser photocoagulation within 30 days prior to surgery day.
* Any type of eye inflammation
* Any punctum inflammation or dacryocystitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-08-07 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
To measure the effect of 0.4mg dexamethasone intracanalicular insert in preventing PME in diabetic patients undergoing cataract surgery when compared to topical prednisolone acetate 1% as measure. | 7 days
  Percentage of eyes that developed post-surgical PME in each group measured on fluorescein angiography at Day 7 on Optical Coherence Tomography at Day 7 by a masked grader.
To measure the effect of 0.4mg dexamethasone intracanalicular insert in preventing PME in diabetic patients undergoing cataract surgery when compared to topical prednisolone acetate 1% as measure. | 30 days
  Percentage of eyes that developed post-surgical PME in each group measured on optical coherence tomography at Day 30 by a masked grader.
To measure the effect of 0.4mg dexamethasone intracanalicular insert in preventing PME in diabetic patients undergoing cataract surgery when compared to topical prednisolone acetate 1% as measure. | 60 days
  Percentage of eyes that developed post-surgical PME in each group measured on fluorescein angiography at Day 60 and on optical coherence tomography at Day 60 by a masked grader.

SECONDARY OUTCOMES:
Incidence of central subfield thickness (CST) at Day 7 post op as seen on optical coherence tomography (OCT) | 7days
  Mean central subfield thickness (CST) at Day 7 post op in each group and comparison between groups.
Incidence of central subfield thickness (CST) at Day 7 post op as seen on optical coherence tomography (OCT) | 30 days
  Mean central subfield thickness (CST) at Day 30 post op in each group and comparison between groups.
Incidence of central subfield thickness (CST) at Day 60 post op as seen on optical coherence tomography (OCT) | 60 days
  Mean central subfield thickness (CST) at Day 60 post op in each group and comparison between groups.
To measure the change in CST inflammation outcomes and in diabetic patients as seen on optical coherence tomography (OCT), Dextenza compared to topical prednisolone acetate 1%. | 7 days
  Mean change in CST from Baseline at Day 7, Day 30 and Day 60 and comparison between groups.
To measure the change in CST inflammation outcomes and in diabetic patients as seen on optical coherence tomography (OCT), Dextenza compared to topical prednisolone acetate 1%. | 30 days
  Mean change in CST from Baseline at Day 7, Day 30 and Day 60 and comparison between groups.
To measure the change in CST inflammation outcomes and in diabetic patients as seen on optical coherence tomography (OCT), Dextenza compared to topical prednisolone acetate 1%. | 60 days
  Mean change in CST from Baseline at Day 7, Day 30 and Day 60 and comparison between groups.
To measure the effect of 0.4mg dexamethasone intracanalicular insert in vision in diabetic patients undergoing cataract surgery when compared to topical prednisolone acetate 1%. | 7 days
  Difference of mean ETDRS Best Corrected Visual Acuity (BCVA) between groups at Day 7 post op
To measure the effect of 0.4mg dexamethasone intracanalicular insert in vision in diabetic patients undergoing cataract surgery when compared to topical prednisolone acetate 1%. | 30 days
  Difference of mean ETDRS Best Corrected Visual Acuity (BCVA) between groups at Day 30 post op
To measure the effect of 0.4mg dexamethasone intracanalicular insert in vision in diabetic patients undergoing cataract surgery when compared to topical prednisolone acetate 1%. | 60 days
  Difference of mean ETDRS Best Corrected Visual Acuity (BCVA) between groups at Day 60 post op
Difference patients with absence of anterior chamber (AC) cells at Day 7 post op | 7 days
  Percentage of patients who had absence of Anterior Chamber (AC) cells at Day 7
Difference patients with absence of anterior chamber (AC) cells at Day 30 post op | 30 days
  Percentage of patients who had absence of Anterior Chamber (AC) cells at Day 30
Difference patients with absence of anterior chamber (AC) cells at Day 60 post op | 30 days
  Percentage of patients who had absence of Anterior Chamber (AC) cells at Day 60
Self reported patient experience of comfort | 60 days
  Self-reported patient experience of comfort (right eye vs. left eye) at Day 60.
Rescue Therapy | 60 days
  Percentage of eyes rescued in each group.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Feldman, MD, Principal Investigator — Ophthalmic Consultants of the Capital Region
Locations (1):
- Ophthalmic Consultants of the Capital Region, Troy, New York, United States